CLINICAL TRIAL: NCT00611078
Title: Environmental Pollutants and the Risk of Soft Tissue Sarcoma: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Engel, Lawrence Stuart, PhD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 04-088
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft Tissue Sarcoma; environment; pollutants; 04-088
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, adipose tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the feasibility of conducting a large hospital based case control study of the role of dioxins and dioxinlike polychlorinated dibenzofurans (PCDFs) and polychlorinated biphenyls (PCBs).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Soft tissue sarcoma at MSKCC are eligible for this study if they meet the following criteria:
* Between 18 and 79 years of age
* were diagnosed within the previous 6 months with primary soft tissue sarcoma of one of the following histologic subtypes: liposarcoma, leiomyoscaroma, MFH, or synovial sarcoma
* are enrolled in protocol 02-060 ("Novel Biochemical and Molecularr Determinants for Soft Tissue Sarcoma"; PI, Dr. Samuel Singer)
* controls will be eligibile for this study if they meet the following criteria
* are b/w 18-79 years of age
* have no prior history of cancer (other than non melanoma skin cancer)

Exclusion Criteria:

* Individuals will be excluded if they
* are unable to sign informed consent for medical or other reasons
* do not speak english

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Soft Tissue Sarcoma at Memorial Sloan Kettering Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2004-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
enrollment of 60 participants | Conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Engel, Ph.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States